CLINICAL TRIAL: NCT07254871
Title: A Phase 2, Randomized, Double-Blind, Placebo-controlled Study to Investigate the Safety and Efficacy in Reducing Nasal Allergen Challenge Provoked Symptoms of Treatment With DM-101PX in Adults With Birch Pollen Allergic Rhinitis or Rhinoconjunctivitis
Brief Title: Study of DM-101PX in Adults With Birch Pollen Allergy
Acronym: BASIT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Desentum Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM-101-C-004
Record Dates: First submitted 2025-09-23; First posted 2025-11-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Birch Pollen Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DM-101PX (Experimental): weekly subcutaneous administration of ascending doses of DM-101PX for 10 weeks
  Interventions: Biological: DM-101PX
- Placebo (Placebo Comparator): weekly subcutaneous administration of Placebo for 10 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DM-101PX — subcutaneous injection of DM-101PX
  Arms: DM-101PX
Biological: Placebo — Placebo to match DM-101PX administered subcutaneously
  Arms: Placebo

SUMMARY:
Randomized, double-blind placebo-controlled phase 2 trial with the aim to investigate safety and efficacy of DM-101-PX in reducing allergic symptoms provoked by nasal allergen challenge in birch pollen allergic adults. Expanded access to the study treatment is not available.

DETAILED DESCRIPTION:
The study will be carried out in two study sites located in Canada

ELIGIBILITY:
Inclusion Criteria:

* Participant of either sex and any race, aged 18 to 65 years inclusive.
* Documented clinical history of birch pollen-induced allergic rhinitis or rhinoconjunctivitis with symptoms that interfere with daily activities or sleep and remain bothersome despite the use of relevant symptomatic medication, and have been present over, at least, 2 previous allergy seasons.
* Bet v 1 specific serum IgE ≥ 0.7 kAU/L.
* Positive Skin Prick Test to birch pollen allergen, with a wheal diameter ≥ 5 mm.
* Body weight ≥ 50 kg and body mass index (BMI) within the range 18-35 kg/m2 inclusive.

Exclusion Criteria:

* History or findings on physical examination at screening visit of any significant disease or disorder which, in the opinion of the Investigator, could put the participant at risk because of participation in the study, influence the results of the study or the participant's ability to participate in the study.
* History of significant rhinitis, sinusitis, and/or presence of significant symptoms of respiratory allergy due to regular contact with other allergens, not associated with the birch pollen season, that are expected to coincide or potentially interfere with the study allergen challenge assessments, as assessed by the Investigator.
* History of nasal polyps or other nasal oropharyngeal conditions that in the judgement of the Investigator may interfere with study outcome assessments.
* History of chronic obstructive pulmonary disease requiring regular treatment.
* Current diagnosis of uncontrolled, partially controlled or persistent asthma requiring regular (> 6 weeks per year) maintenance use of inhaled corticosteroids. History of severe asthma during the pollen season. History of asthma deterioration that resulted in emergency treatment or hospitalization in the 12 months before screening, or a life-threatening asthma attack at any time in the past.
* Forced Expiratory Volume in one second (FEV1) < 75% of predicted. History of severe drug allergy, severe angioedema or systemic allergic reaction of Grade 3 or greater, according to the World Allergy Organization (WAO) scale, due to any cause.
* History of intolerance to the Investigational Product, rescue medications used for systemic allergic reactions (i.e., adrenaline, antihistamine, glucocorticoids, and beta-2 agonists such as salbutamol), or their excipients.
* History of acute hypersensitivity and/or anaphylaxis to protein therapeutics or components of formulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score (TNSS) after treatment | From baseline to 3 weeks after the last dose
  Change in AUC for TNSS from baseline to post-treatment visit. TNSS is a symptom score consisting of 4 nasal symptoms, each symptom is rated as follows: 0 (none), 1 (mild), 2 (moderate), 3 (severe). TNSS score can very between 0-12.

SECONDARY OUTCOMES:
Adverse events (AEs) | from the start of treatment to 3 weeks after the last dose
  Incidence and characteristics of AEs from the start of treatment to the post-treatment NAC visit.
Laboratory safety evaluations | from the start of treatment to 3 weeks after the last dose
  Number and percentage of participants with new onsets of clinically significant abnormalities (as assessed by the investigator) in laboratory safety evaluations
Vital signs | From the start of treatment to 3 weeks after the last dose
  Number and percentage of participants with new onsets of clinically significant abnormalities (as assessed by the investigator) in vital signs
Adverse Events of Special Interest (AESIs) | From the start of treatment to 3 weeks after the last dose
  Incidence and characteristics AESIs: local injection site reactions and systemic allergic reactions
Change in TNSS after follow-up period | from baseline to 20-30 weeks after the last dose
  Change in AUC for TNSS from baseline to follow-up visit.
Change in Total Symptom Score (TSS) | From baseline to 1) 3 weeks, 2) 20-30 weeks after the last dose
  Change in AUC for TSS from baseline to 1) post-treatment, 2) follow-up visit
Change in Peak Nasal Inspiratory Flow (PNIF) | from baseline to 1) 3 weeks, 2) 20-30 weeks after the last dose
  Change in AUC for PNIF from baseline to 1) post-treatment visit, 2) follow-up visit
Change in blood allergy biomarker levels | From baseline to the 7th injection, the 10th injection, 3 weeks after the last dose, and 20-30 weeks after the last dose.
  Change from baseline to the 7th injection, the 10th injection, post-treatment and follow-up visit in the levels of Bet v 1-specific IgE, IgG1 and IgG4.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Opstelten, PhD, Study Director — Desentum Oy
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie publicly available results will be considered for sharing
  Anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant reidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anonymized participant data will be considered for sharing once the product and indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant reidentification.
Access Criteria: Qualified researchers may request access to patient level data and related study documents: patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants after Desentum has received marketing authorization from major health authorities (e.g. FDA, EMA), has the legal authority to share the data, and has made the study results publicly available.